CLINICAL TRIAL: NCT06914804
Title: Stomasense: A New Route to the Proactive Detection and Management of Leaks Within Ostomy Pouches
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: UUREC/24/0074; MR W029561 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2025-03-26; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Ileostomy - Stoma
Keywords: Ileostomy; Stoma-pouch leakage; peristomal skin; dietary intake; quality of life

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leak detection device (microbutton probes) (Experimental): Leakage events will be detected by microbutton probes, which are attached to the sensing device
  Interventions: Device: Stomasense
- Leak detection device (microwire probes) (Experimental): Leakage events will be detected by microwire probes, which are attached to the sensing device
  Interventions: Device: Stomasense

INTERVENTIONS:
Device: Stomasense — A smart device worn alongside stoma pouch systems which detects onset of a leak.

SUMMARY:
People living with an ileostomy may often experience leaks from their stoma pouches. Leakages are a highly stressful experience, so it is no surprise that worry about leaks is very common among ileostomates and this can contribute to increased anxiety and impact negatively on quality of life. Ileostomates will make changes to their lifestyle to minimise the occurrence of leaks; they may avoid travelling long distances, steer clear of busy social events and often restrict certain food(s) and / or drink(s). The latter stands in the way of achieving a healthy balanced diet and can put ileostomates at risk of developing nutritional deficiencies.

Researchers at ulster university have developed a leak sensor device which can be worn unobtrusively alongside any stoma pouch. The device can detect the early stages of a leak from the stoma bag and alerts the user, meaning they are able to change their pouch before it's too late. Participants will be asked to trial 2 versions of the device, each over a 2-week period. At the beginning and end of each period participants will complete a series of questionnaires to allow the research team to determine device efficacy and impact on quality of life. Food diaries will also be completed by participants to give an indication of how dietary intake can impact the incidence of pouch leakage.

DETAILED DESCRIPTION:
Surgical diversion of the bowel to create an opening in the abdomen (stoma) is a common procedure in the treatment of various gastrointestinal conditions; 21 000 stomas are created in the UK each year and it is estimated that 176 000 - 205 000 individuals in the UK are living with a stoma. This is a life-changing operation which requires significant physical and psychological adaptation particularly as bowel/bladder content is collected in a disposable pouch that adheres to the abdomen. Leakage, especially in public, is a constant worry resulting in decreased social interactions, increased anxiety and depression and can have a tremendous impact on family and work life. The extent of the problem was confirmed by the Ostomy Life Study (2015) which surveyed some 4000 ostomates from 11 different countries and found the majority (91%) of participants reported that leakage of the pouch was a concern with 69% confirming that it was their prime worry and greatly impacted on their quality of life (QoL). Leakage events are very traumatic emotionally and will impact an individual's practical management of their ostomy; stoma effluent in contact with the epidermal layer is a major contributing factor in the development of peristomal skin complications (PCS), this in turn can cause difficulty in adhesion of the baseplate to the affected skin, therefore further contributing to the future leaks.

To put an end to this cycle of worsening skin integrity and subsequent increased frequency of leaks, new leak sensor technology has been developed by Ulster University which can be used with any stoma pouch system to detect the early onset of stoma pouch failure - providing an alert that allows the patient to replace the pouch before catastrophic seepage of bowel/bladder content.

Whilst this new leak sensor technology will be extremely useful in the early detection of leaks, it is important to also consider how an individual's management of their stoma, as well as health and lifestyle behaviours, could be manipulated to further reduce the incidence of leaks and improve QoL. In a previous study, participants identified food consumption (i.e., eating certain foods) as being the most prominent contributor to the incidence of leaks. It has been reported that fruit and vegetables are avoided by ostomates - in particular those with an ileostomy - to help minimise the risk of leaks. Obviously, this is less than ideal, considering the well-established health benefits of consuming a diet rich in fruit and vegetables. At present, there is no evidence confirming the efficacy of restricting dietary intake to reduce the frequency of leaks. Therefore, it is possible that people living with a stoma are unnecessarily restricting their dietary intake and putting themselves at risk of various nutrient deficiencies and associated health conditions.

The over-riding aim of the current proposal is to validate a smart device that can be worn unobtrusively alongside existing stoma pouch systems whilst monitoring the condition of the adhesive skin wafer, such that erosion of the bond can be detected before a leak occurs. This would enable the wearer to replace the pouch avoiding the consequences of leakage and accompanying distress, therefore improving QoL and psychological well-being. The impact of the device on participant well-being will be assessed using a series of validated questionnaires. The sensor is not a medical device as it only interacts with the stoma bag and flange and does not interact directly with the participant or their bodily fluids.

The sensing device will:

1. Accurately detect the onset of leaks.
2. Provide a discrete personal alert (vibration).
3. Allow for wireless connectivity for those requiring carer / nursing support.
4. Allow for differences in patient dexterity; two distinct probe systems (microbutton or microwire sensor) will be validated.

Therefore, this study seeks to test the sensor technology with ileostomates in a cross over study involving microbutton and microwire sensors. This study hopes to achieve an 85% success rate in the accurate detection of leaks.

The secondary aim of this study is to determine associations between dietary intake and the incidence of leakages. This information will have the potential to inform the development of dietary guidelines for those living with a stoma, and to therefore improve overall nutritional status and health of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Living with an ileostomy
* ≥1.5-years post-operative
* Aged 18+ years
* Experiencing frequent leaks (i.e., more than once per week)
* Males and females (not currently pregnant/lactating)
* Self-manging their own stoma
* Access to computer / mobile device for survey completion
* No learning or other disabilities
* Have never used / trialled other leak detection systems

Exclusion Criteria:

* Never had an ileostomy,
* Individuals with previous ileostomy or ostomy (colostomy or urostomy)
* <1.5-year post-operative
* <18 years
* Do not experience frequent leaks (i.e., less than once per week)
* Adults with learning or other disabilities
* Have previously used other leak detection systems
* Pregnant/lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychiatric morbidity | Comparison between treatments over a 2-week period.
  Psychiatric morbidity will be assessed at the beginning and end of each test period using the General Health Questionnaire (GHQ-12).
Psychological well-being | Comparison between treatments over a 2-week period.
  Psychological well-being will be assessed at the beginning and end of each test period using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
General quality of life | Comparison between treatments over a 2-week period.
  General quality of life will be assessed at the beginning and end of each test period using the European Organization for Research and Treatment of Cancer (EORTC) QoL questionnaire for colorectal cancer (EORTCQLQ-CR38).
General quality of life | Comparison between treatments over a 2-week period.
  General quality of life will be assessed at the beginning and end of each test period using the The World Health Organization Quality of Life - BREF (WHOQOL-BREF).
Stress and coping | Change over 2 weeks comparison between treatments
  Stress and coping will be assessed at the beginning and end of each test period using the Perceived Stress Scale (PSS), which is a global measure of stress
Resillience | Change over 2 weeks comparison between treatments
  Resillience will be assessed at the beginning and end of each test period using the Connor-Davidson Resilience Scale (CD-RISC)
Stoma related quality of life | Comparison between treatments over a 2-week period.
  Stoma related quality of life will be assessed at the beginning and end of each test period using the Stoma QoL: A Quality-of-Life Questionnaire for People with an Ostomy

SECONDARY OUTCOMES:
Device accuracy | Measured over 2 weeks comparison between treatments
  Participants will keep a daily leak diary in which the incidence of leaks will be recorded. Participants will log leakage events as true positive (TP; successful detection of leak), false positive (FP; sensor alert but no leak occurred) or false negative (FN; occurrence of leak but no alert from device).
Device usability | Measured at 2 weeks comparison between treatments
  Participants will complete a user experience survey at the end of each treatment period.
Dietary intake | Measured over 2 weeks comparison between treatments
  Participants will complete 4-day food diaries at the beginning and end of each treatment period.
Peristomal skin condition | Comparison between treatments over a 2-week period.
  Participants will complete a short questionnaire which evaluates peristomal skin condition at the beginning and end of each treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ulster University, Human Intervention Studies Unit, Coleraine, Co. Derry, United Kingdom

IPD SHARING:
Plan to Share IPD: No